CLINICAL TRIAL: NCT00444795
Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Sutene
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181146
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: SUTENE; post-marketing surveillance; GIST; RCC; Korea
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients diagnosed as GIST after disease progression on or intolerance to imatinib mesylate
  Interventions: Drug: Sunitinib malate
- 2: patients diagnosed as advanced RCC
  Interventions: Drug: Sunitinib malate
- 3: patients diagnosed as unresectable, well-differentiated advanced and/or metastatic pancreatic neuroendocrine carcinoma
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib : dosing not pre-determined
  Groups: 1
Drug: Sunitinib malate — Sunitinib : dosing not pre-determined
  Groups: 2
Drug: sunitinib malate — Sunitinib : dosing not pre-determined
  Groups: 3

SUMMARY:
To monitor use in real practice including adverse events and efficacy on Sutent capsules (Sunitinib malate)

DETAILED DESCRIPTION:
All the patients prescribed according to approved indications at contracted institutions

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as gastrointestinal stromal tumor (GIST) after disease progression on or intolerance to imatinib mesylate, or advanced renal cell carcinoma (aRCC) will be included in the study, or patients diagnosed as unresectable, well-differentiated advanced and/or metastatic pancreatic neuroendocrine carcinoma.

Exclusion Criteria:

* Any patient who does not agree that Pfizer and companies working with Pfizer use his/her information will be excluded.
* Patients with hypersensitivity to sunitinib malate or to any other component of Sutent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed as GIST after disease progression on or intolerance to imatinib mesylate or patients diagnosed as advanced RCC or patients diagnosed as unresectable, well-differentiated advanced and/or metastatic pancreatic neuroendocrine carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2007-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- South Korea (46):
  - Keimyung University Dongsan Medical Center, Jung-gu, Daegu
  - Daegu Catholic University Medical Center, Nam-gu, Daegu
  - GangNeung Asan Hospital, Gangneung-si, Gangwon-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital (SNUH), Seoul, Seoul
  - Hwasun Hospital, Chonnam National University, Cheonnam, South Jeolla Province
  - Hallym University Sacred Heart Hospital, Anyang
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Dong-A University Hospital, Busan
  - Dong-A University Medical Center (Dong-A University Hospital), Busan
  - Dong-A University Medical Center, Department of Medicine, Division of Hemato-Oncology, Busan
  - Hwasun Hospital, Chonnam National University, Cheonnam
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Medical Center, Daegu
  - Daegu Catholic University Medical Center (DCUMC), Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - Chosun University Hospital, Gwang Joo
  - Pusan National University Hospital, Gyeongsangnam-do
  - Wonkwang University School of Medicine and Hospital (WUH), Iksan -Si
  - Inha University Hospital, Incheon
  - Gachon University Gil Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Yeungnam University Medical Center, Nam-gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Medical Center, Seoul
  - KyungHee University Medical Center, Seoul
  - Samsung Medical Center, Dept. of Medicine, Div. of Hematology/Oncology, Seoul
  - Samsung Medical Center/Division of Hematology-Oncology, Department of Medicine, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center/Department of Oncology, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul ST. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju College of Medicine, Wonju Christian Hospital, Wŏnju

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181146&StudyName=Post%20Marketing%20Surveillance%20Study%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Sutene

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This post marketing surveillance (PMS) study enrolled 520 participants between December 2007 and March 2015. Data from 100 participants were obtained from a previously completed study (A6181037).
Groups:
- Sutene: Participants were administered with Sutene as part of routine clinical practice. The use and dosage recommendations for Sutene were based on the approved local product document and were adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Sutene
Started | 620
Completed | 617 (Refer to the Safety Analysis Set.)
Not Completed | 3
Not completed — Not Treated | 1
Not completed — Treated Prior to the Contract Date | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who administered Sutene at least once and were evaluated upon its related safety endpoints at least once.
Arm/Group | Sutene
Number analyzed (Participants) | 617
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.94 (11.29)
Gender [Count of Participants; unit: Participants]
  Female | 149
  Male | 468
Diagnosis [Number; unit: Participants]
  Advanced Renal Cell Carcinoma | 550
  Gastrointestinal Stromal Tumor | 64
  Progressive Pancreatic Neuroendocrine Carcinoma | 2
  Data Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)/Adverse Drug Reactions (ADRs), Serious AEs (SAEs)/Serious ADRs (SADRs), Unexpected AEs/ADRs, and Unexpected SAEs/SADRs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have had a causal relationship with the treatment or usage. All AEs reported after the start of administration of Sutene were considered as treatment-emergent and summarized. All AEs, except for those with causal relationship to the study drug assessed as "unlikely" or "no" (for data that came from Study A6181037), were considered as ADRs. Unexpected AEs/ADRs were classified by medical review with reference to the local product document and confirmed by Pfizer.
Time Frame: From the time that the participant signed data privacy statement through and including 28 calendar days after the last administration of the study drug, average of 27.2 weeks.
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sutene
Number analyzed (Participants) | 617
Percentage of Participants
  AEs | 80.23 [77.08 to 83.37]
  ADRs | 76.50 [73.15 to 79.85]
  SAEs | 11.67 [9.14 to 14.20]
  SADRs | 7.46 [5.39 to 9.53]
  Unexpected AEs | 44.57 [40.65 to 48.49]
  Unexpected ADRs | 35.17 [31.40 to 38.94]
  Unexpected SAEs | 6.32 [4.40 to 8.24]
  Unexpected SADRs | 2.76 [1.47 to 4.05]

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: The antitumor efficacy was measured by objective tumor assessments according to the RECIST of uni-dimensional evaluation. CR was defined as disappearance of all target and non-target lesions, and no new lesions. PR was defined as disappearance of all target lesions, a persistence of ≥1 non-target lesions, no new lesions; or a ≥30% decrease in the sum of the longest dimensions of the target lesions, no unequivocal progression of existing nontarget lesions, no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), no unequivocal progression of existing non-target lesions, and no new lesions. PD was defined as a ≥20% increase in the sum of the longest dimensions of the target lesions; or unequivocal progression of existing non-target lesions, or the appearance of ≥1 new lesions.
Time Frame: At the end of study treatment, average of 23.2 weeks.
Population: Intent-to-treat Analysis Set: Participants who administered Sutene at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sutene
Number analyzed (Participants) | 515
Percentage of Participants | 77.48 [73.87 to 81.08]

ADVERSE EVENTS:
Time Frame: From the time that the participant signed data privacy statement through and including 28 calendar days after the last administration of the study drug, average of 27.2 weeks.
Description: The same event may appear as both an AE and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sutene
Serious Adverse Events (participants affected / at risk) | 72/617
Other Adverse Events (participants affected / at risk) | 474/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sutene (N=617)
Anorexia (Nervous system disorders) | 1
Ascites (General disorders) | 1
Asthenia (General disorders) | 14
Condition aggravated (General disorders) | 5
Death (General disorders) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Oedema (General disorders) | 1
Pain (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiomegaly (Cardiac disorders) | 1
Circulatory failure (Vascular disorders) | 2
Congestive heart failure (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Convulsions (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
hypothyroidism (Endocrine disorders) | 1
Abdomen enlarged (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Appendicitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhage rectum (Gastrointestinal disorders) | 1
Hiccup (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal fistula (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Bilirubinaemia (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Carcinoma of oesophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Purpura thrombopenic thrombotic (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental deficiency (Psychiatric disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Haemolytic-uraemic syndrome (Blood and lymphatic system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8
Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Shock septic (Vascular disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 2
Laceration (Injury, poisoning and procedural complications) | 1
Post-operative wound infection (Injury, poisoning and procedural complications) | 1
Surgical intervention (Surgical and medical procedures) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 5
Urinary tract infection (Renal and urinary disorders) | 2
Haemorrhage intracranial (Vascular disorders) | 1
Haemorrhage nos (Vascular disorders) | 1
Thromboembolism (Vascular disorders) | 1
Thrombophlebitis deep (Vascular disorders) | 1
Conjunctivitis (Eye disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sutene (N=617)
Anorexia (Nervous system disorders) | 159
Asthenia (General disorders) | 82
Chest pain (General disorders) | 34
Face oedema (General disorders) | 82
Fatigue (General disorders) | 109
Fever (General disorders) | 32
Oedema (General disorders) | 38
Oedema periorbital (General disorders) | 45
Palmar-plantar erythrodysaesthesia (General disorders) | 191
Hypertension (Vascular disorders) | 59
Dizziness (Nervous system disorders) | 31
Headache (Nervous system disorders) | 50
Hypothyroidism (Endocrine disorders) | 44
Abdominal pain (Gastrointestinal disorders) | 95
Constipation (Gastrointestinal disorders) | 50
Diarrhoea (Gastrointestinal disorders) | 137
Dyspepsia (Gastrointestinal disorders) | 66
Mucositis nos (Gastrointestinal disorders) | 115
Nausea (Gastrointestinal disorders) | 92
Stomatitis (Gastrointestinal disorders) | 145
Vomiting (Gastrointestinal disorders) | 64
Jaundice (Hepatobiliary disorders) | 72
Serum glutamic-oxaloacetic transaminase increased (Hepatobiliary disorders) | 44
Serum glutamate pyruvate transaminase increased (Hepatobiliary disorders) | 32
Back pain (Musculoskeletal and connective tissue disorders) | 67
Myalgia (Musculoskeletal and connective tissue disorders) | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 137
Coughing (Respiratory, thoracic and mediastinal disorders) | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 44
Rash (Skin and subcutaneous tissue disorders) | 80
Azotaemia (Renal and urinary disorders) | 35
Granulocytopenia (Blood and lymphatic system disorders) | 113
Leucopenia (Blood and lymphatic system disorders) | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days